CLINICAL TRIAL: NCT05156021
Title: A Study on the Treatment Strategy of Neovascular Glaucoma Secondary to Proliferative Diabetic Retinopathy
Brief Title: A Study on the Treatment Strategy of NVG Secondary to PDR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RuijinHospital
Record Dates: First submitted 2021-10-14; First posted 2021-12-14 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2021-10

CONDITIONS: Neovascular Glaucoma; Proliferative Diabetic Retinopathy
MeSH Terms: conditions — Glaucoma, Neovascular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pre-vitrectomy anti-VEGF injection group (Experimental): Patient in this group receive an intravitreal injection of anti-VEGF drug 3-5 days before surgery, followed by PPV combined with PRP and pressure-reducing valve implantation
  Interventions: Drug: anti-VEGF
- pre and post-vitrectomy anti-VEGF injection group (Experimental): Patient in this group receive two intravitreal injections of anti-VEGF drugs. One is injected 3-5 days before surgery, the other is at the same time as the PPV combined with PRP and pressure reducing valve implantation is completed.
  Interventions: Drug: anti-VEGF

INTERVENTIONS:
Drug: anti-VEGF — To explore whether adding post-vitrectomy anti-VEGF agent injection can reach a better prognosis in PDR patients with NVG who underwent PPV combined with PRP and pressure-reducing valve implantation

SUMMARY:
With the increasing incidence of proliferative diabetic retinopathy (PDR), subsequent neovascular glaucoma (NVG) has become one of the main causes of blindness in PDR patients, and the intraocular pressure of PDR patients with NVG is often stubborn. For these patients, not only is the effect of drugs in lowering intraocular pressure poor, but the results of surgery are often unsatisfactory. Because of its poor prognosis, clinical research for better strategy is of great significance in the current situation. At present, for such patients, a combination of effective control of intraocular pressure and treatment of the primary disease is often used. The purpose of this study was to investigate the clinical effects of preoperative with/without intraoperative anti-vascular endothelial growth factor (VEGF) drug therapy combined with pars plana vitrectomy (PPV), pan-retinal photocoagulation (PRP), and pressure-reducing valve implantation in patients with NVG secondary to PDR. Furthermore, the changes of neurotrophic factors in the vitreous humor before and after anti-VEGF treatment will be explored.

ELIGIBILITY:
Inclusion Criteria:

* male or female patients aged over 18 years diagnosed with type 1 or 2 diabetic mellitus (DM) confirmed by experienced endocrinologists. Active PDR and NVG was clinically evident across these patients. The indications to perform surgery included vitreous hemorrhage or fibrous proliferation in the macular area, together with uncontrolled intraocular pressure.

Exclusion Criteria:

* (i) coexistent ocular disease that may interfere with visual outcome; (ii) previous history of vitrectomy or anti-VEGF pharmacotherapy in either eye; (iii) a macula-involving retinal detachment for >6 months in the study eye; (iv) severe external ocular infection; (v) usage of anticoagulant or antiplatelet therapy; (vi) preoperative or postoperative poor diabetes control [serum hemoglobin A1c (HbA1c) >11.0%]; (vii) uncontrolled systemic diseases, such as hypertension, cardiac diseases or presenting abnormal coagulation-associated blood diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2021-12-12 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in Best Corrected Visual Acuity from baseline to 12 months after surgery | Follow-up on the first day, first week, 1, 3, 6, 9 and 12 months after surgery
Changes in Intraocular Pressure from baseline to 12 months after surgery | Follow-up on the first day, first week, 1, 3, 6, 9 and 12 months after surgery

SECONDARY OUTCOMES:
Changes in Neovascularization Recurrence Rate from baseline to 12 months after surgery | Follow-up on the first day, first week, 1, 3, 6, 9 and 12 months after surgery
Changes in Ocular and Systemic Adverse Events from baseline to 12 months after surgery | Follow-up on the first day, first week, 1, 3, 6, 9 and 12 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Xi Shen, Principal Investigator — Ruijin Hospital, Affiliated Shanghai Jiaotong University School of Medicine
Locations (1):
- Ruijin Hospital Affiliated to Shanghai Jiaotong University School of Medicine,, Shanghai, China

IPD SHARING:
Plan to Share IPD: No